CLINICAL TRIAL: NCT04002609
Title: The Systemic and Brain Oxygen Stauration Change During Bronchoscopy
Acronym: BFNIRS
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, Head, Division of General, Vascular and Thoracic Anesthesia, University of Debrecen
Other Study IDs: DE KK RKEB/IKEB 4989-2018; 29215/2017 (Registry Identifier: Government Offices Public Health Administration Organization); DE KK RKEB/IKEB 4989-2018 (Registry Identifier: Local Ethic Comittee University of Debrecen)
Record Dates: First submitted 2019-06-18; First posted 2019-06-28 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: NIRS
Keywords: bronchoscopy, NIRS
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A, Active comparator: Patients in this group did not receive any rountine oxygen supplementation during the procedure. Rescue supplemental oxygen through nasal cannual was provided if clinically significant desaturation could be observed during bronchoscopy. This significant desaturation was defined as systemic oxygen saturation ≤90% on pulsoxymetry or a relative change of ≥ 4% lasting for 1 minute. N=31 patients
- Group B, Active comparator: Supplemental oxygen was provided for the patients through nasal cannula by a flow rate of 2 l/minutes throughout the procedure. N= 31 patients
  Interventions: Other: oxygen
- Group C, Active comparator: Supplemental oxygen administration through nasal cannula by a flow rate of 4 l/minutes throughout the procedure. N= 30 patients
  Interventions: Other: oxygen

INTERVENTIONS:
Other: oxygen — oxygen supplementation during brronchoscopy
  Groups: Group B, Active comparator; Group C, Active comparator

SUMMARY:
Bronchofiberoscopy is a widespread invasive intervention in clinical practice with a number of diagnostic and therapeutic indications. The Clinic of Pulmonary Medicine in Debrecen carries out nearly 2000 examinations a year. The intervention is guided by the recommendation of the Vocational College for Pulmonary Medicine in 2005, but it does not contain a clear recommendation on the oxygen therapy used during the intervention. The Hungarian recommendation states that pulsoximetry is mandatory in bronchoscopy, but it does not contain information on the indications and the implementation of oxygen suplementation. The British Thoracic Society Guideline 2013 deals with the issue and makes the following statements:

* patients should be monitored for oxygen saturation under bronchofiberoscopy
* oxygen supplementation during the test is recommended if the patient's desaturation is significant (greater than 4% or less than 90%) and is over 1 minute
* during the bronchoscopy, the occurrence of oxygen saturation decreases depending on the level of initial oxygen saturation, respiratory function, co-morbidity, sedation and the course of intervention.

The aim of our study is to investigate the frequency with which systemic hypoxia occurs during bronchoscopy, what factors may contribute to its development and how the level of cerebral oxygen saturation changes with systemic desaturation (in the case of NIRS, a 20% reduction from baseline is considered significant).

DETAILED DESCRIPTION:
: Consecutive patients admitted to Bronchology Laboratory of Department of Pulmonology, University of Debrecen for flexible bronchoscopy were asked to participate in the study. After explaining the procedure in detail, all patients gave written informed consent.

The indication of flexible bronchoscopy was based in all cases on the results of medical history, physical examination, chest X-ray and/or chest CT scan, lung function tests and laboratory parameters including hemoglobin concentration, hemostasis variables as well as blood gas analysis when necessary.

Bronchoscopy (PENTAX EB-1975K) was performed after an at least 4-hour fasting period. The procedure was performed either in sitting or supine position after a topical administration of lidocaine 2% solution. Routine monitoring consisted of ECG, non-invasive blood pressure measurement, pulse oxymetry (finger probe). As an additional monitoring tool, near infrared monitoring sensor was placed to the forhead of the dominant hemisphere of patients for monitoring cerebral oxygen saturation. INVOS 5100 C cerebral oximeter (Covidien llc, 15 Hampshire Street, Mansfield, MA 02048 USA) was used for cerebral near infrared spectroscopy measurements.

ELIGIBILITY:
Inclusion Criteria:

inclusion criteria: adult patients (over 18 years) going elective bronchoscopy

Exclusion Criteria:

age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Bronchology Laboratory of Department of Pulmonology, University of Debrecen for flexible bronchoscopy were asked to participate in the study. After explaining the procedure in detail, all patients gave written informed consent.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
systemic oxygen saturation | during bronchoscopy
  measure systemic oxygen saturations with Infinity Delta XL

SECONDARY OUTCOMES:
cerebral oxygen saturation | during bronchoscopy
  measure cerebral oxygen saturation with INVOS Model 5100C Cerebral I Somatic Oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD, DSci, Principal Investigator — Department of Anesthesiology and Intensive Care, University of Debrecen, Health and Medical Science Centre
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasko A, Kovacs S, Fulesdi B, Molnar C. Assessment of Systemic and Cerebral Oxygen Saturation during Diagnostic Bronchoscopy: A Prospective, Randomized Study. Emerg Med Int. 2020 Dec 9;2020:8540350. doi: 10.1155/2020/8540350. eCollection 2020. PMID 33505726